CLINICAL TRIAL: NCT04828395
Title: Fluzoparib Combined With Camrelizumab for Maintenance Treatment of Locally Advanced Non-small Cell Lung Cancer After Concurrent Chemotherapy and Radiotherapy. A Single-arm, Single-center, Phase II Clinical Study
Brief Title: Fluzoparib Combined With Camrelizumab for Maintenance Treatment of Locally Advanced Non-small Cell Lung Cancer
Acronym: F&C
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210094A
Record Dates: First submitted 2021-03-21; First posted 2021-04-02 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; fluzoparib; PE regimen; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Camrelizumab — 200mg iv Q3W
Drug: Fluzoparib — 150mg bid
Drug: Cisplatin，Pemetrexed — Cisplatin 75mg/m2 IV and Pemetrexed 500mg/m2 IV Q3W (Day 1 of each cycle of cycles 1-3) (non-squamous cell carcinoma only)
Drug: Cisplatin，Etoposide — Cisplatin 50mg/m2 IV (the 1st and 8th days of the 1st cycle and the 2nd cycle; the 8th and 15th days of the 3rd cycle); Etoposide 50mg/m2 IV (the 1st cycle And the 1st to the 5th day of the 2nd cycle; the 8th to the 12th day of the 3rd cycle).
Drug: Carboplatin, Albumin Paclitaxel — Carboplatin AUC=6, Albumin Paclitaxel 100mg/m2 IV; Days 1, 8 and 15 of cycles 1, 2, and 3.
Radiation: Radiotherapy — 60 Gy (total 6 weeks)

SUMMARY:
Fluzoparib combined with Camrelizumab for maintenance treatment of locally advanced non-small cell lung cancer after concurrent radiotherapy and chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Subject type and disease characteristics

  1. Suffer from NSCLC diagnosed by pathology (histology or cytology).
  2. Have stage IIIA, IIIB, or IIIC NSCLC diagnosed according to the 8th edition of the American Joint Committee on Cancer.
  3. It is confirmed and recorded by the multidisciplinary oncology committee or the treating physician and the thoracic surgeon to have stage III NSCLC that cannot accept radical surgery.
  4. In whole-body fluorodeoxyglucose (FDG)-PET or FDG-PET/CT and diagnostic-quality CT or MRI scans of the chest, abdomen, pelvis, and brain, there is no evidence of metastatic disease as stage IV NSCLC.

     Note: Unless otherwise proven, the presence of pleural/pericardial effusion is considered to indicate metastatic disease. For the presence of pleural effusion in both the CT chest scan and the chest X-ray in the front view, thoracentesis is required to confirm that the pleural effusion is cytologically negative. Exclude participants whose effusion is exudate, even if the effusion is cytologically negative. Subjects who have met the remaining inclusion/exclusion criteria and whose pleural effusion is not visible on chest X-rays in the front and side views, or who have too little effusion to be safely extracted can enter the study.
  5. Suffer from a measurable disease defined by RECIST 1.1, and at least one lesion is suitable as a target lesion (determined by the investigator/imaging review of the local research center).
  6. No previous treatment (chemotherapy, targeted therapy or radiotherapy) for stage III NSCLC.
  7. A tumor tissue sample (tissue biopsy [thick needle biopsy, excision biopsy, or excision biopsy]) is provided. The tissue block of FFPE is better than the slice. The newly obtained tumor sample is better than archived tissue and should be obtained before chest imaging at screening.

     Note: If an unstained section is submitted, the new section must be submitted to the testing laboratory within 14 days of preparation.
  8. The ECOG performance status assessed within 7 days before the first dose of the study intervention is 0 or 1 point.
  9. The life expectancy is at least 6 months.
  10. Sufficient PFT is defined as FEV1> 50% of predicted normal expiratory volume and lung carbon monoxide diffusion volume (DLCO)> 40% of predicted normal value. For subjects without DLCO measurement values, if the measured pulse oximetry (O2 saturation) in indoor air is ≥90%, it will be deemed to have sufficient oxygen transmission.
  11. Have adequate organ functions, as defined in Table 1; all laboratory tests during the screening period should be completed 10 days before the start of the research intervention.

      1. ANC ≥ 1.5×109/L;
      2. HB ≥ 90 g/L;
      3. PLT ≥ 100×109/L;

      The biochemical inspection must meet the following standards:
      1. TBIL ≤ 1.5ULN;
      2. ALT, AST≤ 2.5 ULN;
      3. Serum creatinine sCr≤1.5ULN, endogenous creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
      4. Coagulation function must meet: INR≤1.5 and APTT≤1.5ULN;
      5. Heart color Doppler ultrasound LVEF≥50% Demographics
  12. Men or women who are at least 18 years old and up to 120 years old (including 18 and 120 years old) when signing the informed consent form.

      Male subjects The contraceptive measures used by men should comply with the local regulations regarding contraceptive measures participating in clinical research.
  13. Male subjects must agree to take contraceptive measures during treatment and at least 180 days after the last dose of the study intervention.

      Note: Male subjects must avoid donating sperm during treatment and for at least 180 days after the last dose of the study intervention.

      Female subjects The contraceptive measures used by women should comply with local regulations regarding contraceptive measures participating in clinical research.
  14. Female subjects who are not pregnant, are not breastfeeding, and meet at least one of the following conditions, can participate in the study:

      1. Women of non-bearing age. or
      2. Agree to take contraceptive measures during treatment and at least 180 days after the administration of the last study intervention Informed consent
  15. Subjects (or their legal representatives, if applicable) provide written informed consent to participate in the study. Subjects may also need to provide informed consent for future biomedical research. However, subjects can only participate in the main experiment and not participate in future biomedical research.

Exclusion Criteria:

* Patients with any of the following cannot be included in this study:

Medical condition

1. People with small cell lung cancer or mixed tumors with small cell components and positive for EGFR, ALK and other driver genes. Note: Subjects with squamous NSCLC are not eligible for chemotherapy with pemetrexed.
2. Have a medical history of MDS/AML, current diagnosis or features suggestive of these diseases.
3. There is a record of weight loss> 10% (from baseline) in the past 3 months. Previous/combined treatment
4. There is a radiotherapy plan in which the whole lung (whole lung V20-GTV) receiving a total dose of >20 Gy (V20) may exceed 34% of the lung volume.

   Note: Subjects must be evaluated by a radiation oncologist during screening.
5. Received previous chest radiotherapy, including radiotherapy for esophagus, mediastinum or breast cancer.
6. Have previously received anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that target another stimulating or co-inhibitory T cell receptor (such as CTLA-4, OX-40, CD137) treatment.
7. Have previously received fluzoparib or any other PARP inhibitor treatment.
8. Underwent major surgery (other than vascular access) within 4 weeks before the first administration of the study drug.

   Note: If the subject has undergone major surgery or vascular access, it must have fully recovered from treatment toxicity and/or complications before starting the research intervention.
9. It is expected that any other form of anti-tumor therapy will be required during the study period.
10. Live vaccines have been vaccinated within 30 days before the first administration of the test drug. Examples of live vaccines include, but are not limited to, the following vaccines: measles, mumps, rubella, varicella/shingles (chickenpox), yellow fever, BCG, and typhoid vaccine. Since seasonal influenza vaccines for injection are usually inactivated virus vaccines, their use is permitted; however, intranasal influenza vaccines (for example, FluMist®) are live attenuated vaccines, so their use is not allowed.
11. Received colony stimulating factor (such as granulocyte colony stimulating factor [GCSF], granulocyte-macrophage colony stimulating factor [GM-CSF] or recombinant erythropoietin) within 28 days before the first administration of the research intervention.
12. Currently receiving strong inducers of CYP3A4 (phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine) that cannot be discontinued during the study period And St. John's Wort) or intermediate inducers (such as bosentan, efavirenz, modafinil). Before starting fluzoparib treatment, pentobarbital needs a washout period of 5 weeks, and other drugs need a washout period of 3 weeks.
13. Currently receiving strong inhibitors of cytochrome P450 (CYP) 3A4 that cannot be discontinued during the study period (such as itraconazole, telithromycin, clarithromycin, boosted with ritonavir or cobiastat) Protease inhibitors, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate inhibitors (such as ciprofloxacin, erythromycin, diltiazem, fluconazole) , Verapamil). The washout period required before initiating fluzoparib is 2 weeks.

    Pemetrexed specific
14. At least 2 days before pemetrexed administration (5 days for long-acting drugs (such as piroxicam)), during administration, and at least 2 days after administration, aspirin or other NSAIDs cannot be suspended, except for the daily dose of aspirin ≤1.3 grams outside.
15. Unable/unwilling to take folic acid, vitamin B12 and dexamethasone. Past/concurrent clinical research experience
16. Are currently participating in or have previously participated in research drug research, or have used research devices within 4 weeks before the first administration of the research intervention.

    Note: Subjects who have entered the follow-up period of the experimental study can participate in this study as long as it is more than 4 weeks after the last administration of the previous investigational drug.

    Diagnostic evaluation
17. According to the investigator's judgment, resting electrocardiogram (ECG) indicates uncontrolled and potentially reversible heart disease (for example, unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, electrolyte imbalance, etc.) , Or the subject has congenital long QT syndrome.
18. Have a diagnosis of immunodeficiency or are receiving chronic systemic steroid therapy (taking more than 10 mg prednisone or equivalent daily) or any form of immunosuppressive therapy within 7 days before the first administration of the study drug.

    Note: The following indications allow the use of glucocorticoids:
    * For eye, intranasal or topical use.
    * Inhalers for the management of asthma or chronic obstructive pulmonary disease.
    * Systemic physiological corticosteroid replacement therapy for hormone replacement therapy, prevention of vomiting, regulation of symptoms suspected of immunological etiology, or as a pretreatment for IV contrast agent allergy or chemotherapeutics.
19. In the past 5 years, there are other malignant tumors that are progressing or require active treatment.

    Note: Patients with skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder that have received potential radical treatment Subjects with cystic carcinoma or carcinoma in situ (eg, breast cancer, cervical cancer in situ) may not be excluded.
20. Severely allergic to research intervention and/or any of its excipients (≥Grade 3).
21. Suffered from an active autoimmune disease that requires systemic treatment in the past 2 years (ie use of disease modifiers, corticosteroids, or immunosuppressive agents). Replacement therapies (for example, thyroxine, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) are not considered systemic treatments and are allowed.
22. A history of (non-infectious) pneumonia/interstitial lung disease that requires steroid treatment, or current non-infectious pneumonia/interstitial lung disease. Lymphatic spread of NSCLC is not an exclusion criterion.
23. Have an active infection that requires systemic treatment.
24. Known history of human immunodeficiency virus (HIV) infection. Unless mandatory by local health authorities, HIV testing is not required.
25. A known history of hepatitis B (defined as HBsAg responsiveness) or active hepatitis C virus (defined as detection of HCV RNA [qualitative]) infection.

    Note: Hepatitis B and C tests are not required unless required by local health authorities
26. Patients with active tuberculosis (TB; Mycobacterium tuberculosis) and are being treated (unless mandatory by the local health authority, TB testing is not required; subjects who have received previous treatment are allowed to enter the group).
27. There is historical or current evidence of any disease, treatment, or abnormal laboratory value that may interfere with the results of the research, prevent the subject from participating in the research throughout, or cause the researcher to believe that participating in the research is not in the subject's best interests.
28. According to the opinions of treatment investigators, serious, uncontrolled medical diseases or non-malignant systemic diseases are regarded as adverse medical risks. Examples include, but are not limited to: uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled grand mal seizures, unstable spinal cord compression, or superior vena cava syndrome.
29. Suffer from known mental illness or substance abuse disease, and these diseases will interfere with the subject's ability to cooperate with the research requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review | 2 year
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review | 2 year
  ORR is defined as the percentage of participants who have achieved a Complete Response (CR) or a Partial Response (PR)
Disease control rate (DCR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review | 2 year
  Disease control rate is the proportion of patients whose tumors have shrunk or stabilized for a certain period of time, including complete remission (CR), partial remission (PR) and stable (SD) cases
Overall Survival (OS) | 2 year
  OS was defined as the time from randomization to death due to any cause. OS is presented. Censoring will be performed using the date of last known contact for those who are alive at the time of analysis.
Safety of drug application | 2 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Liu ningbo, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided